CLINICAL TRIAL: NCT01380210
Title: MRI Findings of Encephalopathy Associated With Carbon Dioxide (CO2) Intoxication
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: China Medical University Hospital, China Medical University Hospital
Other Study IDs: DMR100-IRB-012
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: CO2 Intoxication
Keywords: Carbon dioxide intoxication; Diffusion weighted images(DWI)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Carbon dioxide intoxication is a rare condition and only few case reports are found in the literature. There were six patients who suffered from carbon dioxide intoxication in our hospital about two years ago. Two of them are more severe with conscious change and brain MRI studies of the two patients were performed. Reviewing the literature, no any report has mentioned about the encephalopathy associated with carbon dioxide intoxication. We want to review the brain lesions on the diffusion weighted images and the laboratory data of the patients for further diagnostic help.

ELIGIBILITY:
Inclusion Criteria:

* CO2 intoxication

Exclusion Criteria:

* None CO2 intoxication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-02